CLINICAL TRIAL: NCT03963661
Title: Investigating a Portable Patient-led Virtual Reality Platform for Assessment and Rehabilitation of Hemispatial Neglect: a Usability Study
Brief Title: Investigating Usability of c-SIGHT in the Homes of Brain Injury Survivors
Acronym: c-SIGHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of East Anglia (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Stephanie Rossit, Principal Investigator, University of East Anglia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R206721
Record Dates: First submitted 2019-05-20; First posted 2019-05-28 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Stroke; Brain Injuries; Spatial Neglect; Attention Deficit
Keywords: Telerehabilitation; Spatial neglect; SIGHT; Computorized therapy; Stroke; Innatention; Self-admnistered therapy; Usability
MeSH Terms: conditions — Stroke; Brain Injuries; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- c-SIGHT (Experimental): SIGHT requires participants to grasp and lift rods with their less impaired arm.
  Interventions: Behavioral: c-SIGHT (computorized spatial innatention grasping home-based therapy)

INTERVENTIONS:
Behavioral: c-SIGHT (computorized spatial innatention grasping home-based therapy) — C-SIGHT will be self-administered at people's homes. c-SIGHT is a computerized therapy administered via people's television. The therapy involves performing repeated rod lifts with the less impaired arm in response to auditory and visual instructions presented on the television screen connected to a laptop. A small motion-tracking camera monitors rod lifts during therapy sessions. People will be asked to self-administer c-SIGHT for 1 hour a day (30min after breakfast and 30min after lunch) for 7 consecutive days. The first day of therapy will be performed with a therapist there for training purposes.
  Other Names: visuomotor feedback training

SUMMARY:
A brain injury can damage the brain, so that it no longer receives information about the space around one side of the world. If this happens, people may not be aware of anything on one side, usually the same side they also lost their movement (the most affected side). This severe condition is called spatial neglect. Currently there is no recommended diagnostic test or clinically-proven treatment for the condition. In a recent study, the investigators found a long-lasting reduction in neglect if people practiced picking-up an object with their unaffected hand. This intervention is called Spatial Inattention Grasping Home-based Therapy (SIGHT). It requires people to lift wooden rods of different lengths. Once a person is familiar with the task, they can practice on their own at a time convenient to them in their homes. The investigators have developed the first computerized version of SIGHT (c-SIGHT) as well as a novel diagnostic test for neglect using portable low-cost motion-tracking technology that can be used in the patient's home. In the proposed study, the investigators will investigate how usable and acceptable this technology is in people's homes. Stroke survivors (recruited from community settings) will undergo a 7-day self-led training at their homes with c-SIGHT. At the end of the intervention, 1:1 semi-structured interviews will be carried out with both stroke survivors and carers to investigate usability and acceptability of c-SIGHT. Moreover, spatial neglect, carer burden and motor function will be assessed pre- and post-completion of c-SIGHT.

ELIGIBILITY:
Inclusion Criteria:

* +18
* suffered brain injury
* have TV with around 2 meters in front of it to be able to run the therapy
* live in the Norfolk, Suffolk, Essex or Cambridgeshire (UK)
* no other pre-existing neurological disorders (such as dementia)
* no language impairment (able to follow 1-stage command)
* mental capacity to consent
* no known learning disability
* no major psychiatric illness
* no history of substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-04-03 (Estimated)

PRIMARY OUTCOMES:
Behavioral Inattention Test (BIT) conventional sub tests | Change from baseline (T0) to 7 days (pre-treatment baseline, T1) and from T1 to immediately after 7 days of therapy (T2)
  Standardized measure of spatial inattention

SECONDARY OUTCOMES:
Line bisection Test | Change from baseline (T0) to 7 days (pre-treatment baseline, T1) and from T1 to immediately after 7 days of therapy (T2)
  Test for spatial inattention which measures spatial biases when marking middle of 10 20mm lines. Bisection error bigger that 6mm is considered evidence of spatial inattention.
Broken Hearts test from Oxford Cognitive Screening (paper version) | Change from baseline (T0) to 7 days (pre-treatment baseline, T1) and from T1 to immediately after 7 days of therapy (T2)
  Standardized measure of spatial inattention
Computerized extrapersonal neglect test (CENT) | Change from baseline (T0) to 7 days (pre-treatment baseline, T1) and from T1 to immediately after 7 days of therapy (T2)
  Computerized test measuring ego and allocentric neglect sub types in extra personal space via television screen
Catherine Bergego Scale | Change from baseline (T0) to 7 days (pre-treatment baseline, T1) and from T1 to immediately after 7 days of therapy (T2)
  Standardized checklist to detect presence and degree of unilateral neglect during observation of everyday life situations. The scale also measures self-awareness of behavioral neglect (anosognosia).
  The CBS uses a 4-point rating scale to indicate the severity of neglect for each item:
  0 = no neglect
  1. = mild neglect (patient always explores the right hemispace first and slowly or hesitantly explores the left side)
  2. = moderate neglect (patient demonstrates constant and clear left-sided omissions or collisions)
  3. = severe neglect (patient is only able to explore the right hemispace)
  This results in a total score out of 30.
  Azouvi et al. (2002, 2003) have reported arbitrary ratings of neglect severity according to total scores:
  0 = No behavioral neglect 1-10 = Mild behavioral neglect 11-20 = Moderate behavioral neglect 21-30 = Severe behavioral neglect
Pinch and grip force task (dynamometer) | Change from baseline (T0) to 7 days (pre-treatment baseline, T1) and from T1 to immediately after 7 days of therapy (T2)
  Measures upper limb function
Caregiver Burden Scale | Change from baseline (T0) to 7 days (pre-treatment baseline, T1) and from T1 to immediately after 7 days of therapy (T2)
  To assess perceived burden among people caring for others with disabilities. There are 22 items in which the carer rates perceived burden from 0 (never) to 4 (nearly always).
  A total score of 0 to 20 = little or no burden; 21 to 40 = mild to moderate burden; 41 to 60 = moderate to severe burden; 61 to 88 = severe burden.
Stroke Specific Quality of Life Scale (SS-QOL) | Change from baseline (T0) to 7 days (pre-treatment baseline, T1) and from T1 to immediately after 7 days of therapy (T2)
  A patient-centered outcome measure intended to provide an assessment of health-related quality of life (HRQOL) specific to patients with stroke. Patients must respond to each question of the SS-QOL with reference to the past week. It is a self-report scale containing 49 items in 12 domains. Items are rated on a 5-point Likert scale. Higher scores indicate better functioning. The SS-QOL yields both domain scores and an overall SS-QOL summary score. The domain scores are unweighted averages of the associated items while the summary score is an unweighted average of all twelve domain scores.

OTHER OUTCOMES:
System Usability Scale | immediately after 7 days of therapy (T2)
  To assess usability of devices and applications. Participants are asked to score the following 10 items with one of five responses that range from Strongly Agree to Strongly disagree. The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking.
  Based on research, a SUS score above a 68 would be considered above average and anything below 68 is below average.
Semi-structured interview at end of study with carer and stroke survivor | immediately after 7 days of therapy (T2)
  To assess usability (qualitative data)
WAIS Digit span (control measure) | Change from baseline (T0) to 7 days (pre-treatment baseline, T1) and from T1 to immediately after 7 days of therapy (T2)
  Digit span from WAIS (forward, backward and sequential) is used as a control task

CONTACTS AND LOCATIONS:
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossit S, Benwell CSY, Szymanek L, Learmonth G, McKernan-Ward L, Corrigan E, Muir K, Reeves I, Duncan G, Birschel P, Roberts M, Livingstone K, Jackson H, Castle P, Harvey M. Efficacy of home-based visuomotor feedback training in stroke patients with chronic hemispatial neglect. Neuropsychol Rehabil. 2019 Mar;29(2):251-272. doi: 10.1080/09602011.2016.1273119. Epub 2017 Jan 24. PMID 28116988